CLINICAL TRIAL: NCT01543256
Title: A Multi-Center, Prospective, Randomized Study Comparing Removable, Self-Expanding Metal Stents to Plastic Stents for the Treatment of Benign Biliary Strictures Secondary to Chronic Pancreatitis
Brief Title: WallFlex Biliary Fully Covered (FC) Chronic Pancreatitis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDM00047682
Record Dates: First submitted 2012-02-14; First posted 2012-03-02 (Estimated); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2021-12

CONDITIONS: Biliary Stricture
Keywords: benign biliary strictures secondary to chronic pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metal stents (Active Comparator): The WallFlex Biliary Fully Covered Stent System is being evaluated for treatment of benign biliary strictures secondary to chronic pancreatitis.
  Interventions: Device: WallFlex™ Biliary RX Fully Covered Stent System RMV
- Plastic Stents (Active Comparator): Plastic stents per Investigator preference are being evaluated for treatment of benign biliary strictures secondary to chronic pancreatitis.
  Interventions: Device: Commercially available Plastic Stent Per Investigator preference

INTERVENTIONS:
Device: WallFlex™ Biliary RX Fully Covered Stent System RMV — Temporary placement of the WallFlex Biliary RX Fully Covered Stent for treatment of benign biliary strictures secondary to chronic pancreatitis. The stent will be removed after 12 months indwell. ("RMV" in intervention name indicates "removable")
  Arms: Metal stents
Device: Commercially available Plastic Stent Per Investigator preference — Temporary placement/exchange of multiple biliary plastic stents for treatment of benign biliary strictures secondary to chronic pancreatitis. Stents will be removed after cumulative indwell of 12 months.
  Arms: Plastic Stents

SUMMARY:
The purpose of this of this study is to compare the use of Self Expanding Metal Stents (SEMS) to plastic stents for the treatment of benign biliary strictures secondary to chronic pancreatitis as it pertains to stricture resolution rates, complication rates and number of endoscopic retrograde cholangiopancreatography (ERCP) procedures during 24 months.

Statistical testing will be performed to determine if the rate of stricture resolution for the metal stent is non-inferior to the plastic stent group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Chronic pancreatitis
* Symptomatic bile duct stricture (defined by cholangitis or persistent jaundice for at least one month or cholestasis associated with at least 3 times normal alkaline phosphatase levels) documented at time of enrollment for naïve stricture or at the time of prior plastic stent placement in strictures that had one prior plastic stent inserted.12
* Common bile duct stricture based on imaging assessment of dilatation of the common and/or intrahepatic bile ducts

Exclusion Criteria:

* Biliary stricture of benign etiology other than chronic pancreatitis
* Prior biliary metal stent or any plastic stenting other than one plastic stent of 10 Fr or less for 6 months or fewer
* Developing obstructive biliary symptoms associated with an attack of acute pancreatitis
* Biliary stricture of malignant etiology
* Stricture within 2 cm of common bile duct bifurcation
* Known bile duct fistula or leak
* Subjects for whom endoscopic techniques are contraindicated
* Known sensitivity to any components of the stent or delivery system
* Symptomatic duodenal stenosis (with gastric stasis)
* Participation in another investigational study within 90 days prior to consent
* Investigator Discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-09-18 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D.Nageshwar Reddy, MD, Principal Investigator — Asian Institute of Gastroenterology
Locations (14):
- Australia (2):
  - Royal Prince Alfred Medical Center, Newtown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
- Allgemeines Krankenhaus AKH, Vienna, Austria
- Belgium (2):
  - Erasme Hospital, Brussels
  - UZ Gasthuisberg, Leuven
- CHUM - Hopital Saint-Luc, Montreal, Quebec, Canada
- Hopital Edouard Herriot, Lyon, France
- Evangelisches Krankenhaus Dusseldorf, Düsseldorf, Germany
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Asian Institute of Gastroenterology, Hyderabad, India
- Italy (2):
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona, VR
  - Policlinico Universitario Agostino Gemelli, Rome
- Erasmus Medical Center, Rotterdam, CE, Netherlands
- Karolinska Universitets Sjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Ramchandani M, Lakhtakia S, Costamagna G, Tringali A, Puspoek A, Tribl B, Dolak W, Deviere J, Arvanitakis M, van der Merwe S, Laleman W, Ponchon T, Lepilliez V, Gabbrielli A, Bernardoni L, Bruno MJ, Poley JW, Arnelo U, Lau J, Roy A, Bourke M, Kaffes A, Neuhaus H, Peetermans J, Rousseau M, Reddy DN. Fully Covered Self-Expanding Metal Stent vs Multiple Plastic Stents to Treat Benign Biliary Strictures Secondary to Chronic Pancreatitis: A Multicenter Randomized Trial. Gastroenterology. 2021 Jul;161(1):185-195. doi: 10.1053/j.gastro.2021.03.015. Epub 2021 Mar 17. PMID 33741314

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 172 enrolled participants, 164 met inclusion criteria and were randomized to treatment.
Groups:
- Metal Stents: The WallFlex Biliary Fully Covered Stent System is being evaluated for treatment of benign biliary strictures secondary to chronic pancreatitis.
  WallFlex™ Biliary RX Fully Covered Stent System RMV: Temporary placement of the WallFlex Biliary RX Fully Covered Stent for treatment of benign biliary strictures secondary to chronic pancreatitis. The stent will be removed after 12 months indwell.
Period: Overall Study
Arm/Group | Metal Stents | Plastic Stents
Started | 80 | 84
Completed | 62 | 70
Not Completed | 18 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metal Stents | Plastic Stents | Total
Number analyzed (Participants) | 80 | 84 | 164
Age, Continuous [Median (Full Range); unit: years] | 51 [28 to 74] | 53 [23 to 74] | 52 [26 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 70 | 72 | 142
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 3 | 5
  Netherlands | 5 | 6 | 11
  Austria | 8 | 11 | 19
  Sweden | 3 | 2 | 5
  Belgium | 13 | 13 | 26
  Hong Kong | 2 | 3 | 5
  Italy | 16 | 16 | 32
  Australia | 4 | 3 | 7
  France | 6 | 6 | 12
  Germany | 1 | 1 | 2
  India | 20 | 20 | 40
Time since chronic pancreatitis (CP) diagnosed [Median (Full Range); unit: years] | 3.1 [.1 to 35.8] | 1.7 [.1 to 32.4] | 1.9 [.1 to 35.8]
Gallbladder in situ [Count of Participants; unit: Participants] | 69 | 72 | 141
CP etiology alcoholic [Count of Participants; unit: Participants] — Population: The number of analyzed participants are lower than the overall number of baseline participants because of missing data or status unknown.
  Participants
    number analyzed (Participants) | 71 | 78 | 149
    (all) | 54 | 53 | 107
Calcifying CP [Count of Participants; unit: Participants] — Population: The number of analyzed participants are lower than the overall number of baseline participants because of missing data or status unknown.
  Participants
    number analyzed (Participants) | 74 | 80 | 154
    (all) | 59 | 62 | 121
Candidate for surgery [Count of Participants; unit: Participants] — Population: The number of analyzed participants are lower than the overall number of baseline participants because of missing data or status unknown.
  Participants
    number analyzed (Participants) | 72 | 77 | 149
    (all) | 60 | 61 | 121
Prior plastic stent [Count of Participants; unit: Participants] | 34 | 38 | 72
Prior Biliary Sphincterotomy [Count of Participants; unit: Participants] — Population: The number of analyzed participants are lower than the overall number of baseline participants because of missing data or status unknown.
  Participants
    number analyzed (Participants) | 79 | 82 | 161
    (all) | 39 | 39 | 78
Prior pancreatic sphincterotomy [Count of Participants; unit: Participants] — Population: The number of analyzed participants are lower than the overall number of baseline participants because of missing data or status unknown.
  Participants
    number analyzed (Participants) | 79 | 82 | 161
    (all) | 26 | 27 | 53
Baseline Bilirubin [Median (Full Range); unit: mg/dL] | 1 [.1 to 25.3] | 1.4 [.2 to 17.7] | 1.3 [.1 to 25.3]
Baseline Alkaline Phosphatase [Median (Full Range); unit: IU/L] | 337 [46 to 1871] | 262.5 [55 to 1909] | 299 [46 to 1909]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stricture Resolution
Description: Stricture resolution defined as absence of re-stenting after the 12-month stenting period, and 24 months serum alkaline phosphatase level not exceeding twice the level at the end of stenting period.
Time Frame: After 12-month stenting period through 24 month follow-up (approximately 12 months)
Population: Of 80 participants in metal stent arm, only 62 were eligible for primary endpoint evaluation. Of 84 participants in plastic stent arm, only 70 were eligible for primary endpoint evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Metal Stents | Plastic Stents
Number analyzed (Participants) | 62 | 70
Participants | 47 | 54
Statistical Analysis 1: Comparison: Metal Stents vs Plastic Stents; Test type: Non-Inferiority — Non-Inferiority margin was 20%; p = .008, Exact non-inferiority

2. Secondary Outcome: Serious Adverse Events Related to the Device or Procedure
Description: Device or procedure related serious adverse events from the initial stent placement procedure to the 24 month follow-up.
Time Frame: Initial stent placement procedure to 24 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Metal Stents | Plastic Stents
Number analyzed (Participants) | 80 | 84
Participants | 19 | 16
Statistical Analysis 1: Comparison: Metal Stents vs Plastic Stents; Test type: Superiority; p = .568, Fisher Exact

3. Secondary Outcome: Number of ERCP Procedures Through 24 Months After Initial Stent Placement.
Description: The number of endoscopic retrograde cholangiopancreatography (ERCP) procedures through 24 months, after initial stent placement.
Time Frame: Initial stent placement procedure to 24 month follow-up
Population: Of 80 participants in metal stent arm, 1 participant failed technical success at baseline and did have a completed ERCP procedure. Of 84 participants in plastic stent arm, 2 participants failed technical success at baseline and did have a completed ERCP procedure.
Measure: Mean (Standard Deviation); unit: procedures
Arm/Group | Metal Stents | Plastic Stents
Number analyzed (Participants) | 79 | 82
procedures | 2.6 (1.3) | 3.9 (1.3)
Statistical Analysis 1: Comparison: Metal Stents vs Plastic Stents; Test type: Superiority; p < .001, Negative binomial

4. Secondary Outcome: Ability to Deploy Stent(s) in Satisfactory Position (Technical Success)
Description: Technical success defined as the ability to deploy the stent(s) in satisfactory position during initial stent placement procedure.
Time Frame: Initial stent placement procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Metal Stents | Plastic Stents
Number analyzed (Participants) | 80 | 84
Participants | 79 | 82
Statistical Analysis 1: Comparison: Metal Stents vs Plastic Stents; Test type: Superiority; p = .99, Fisher Exact

5. Secondary Outcome: Length of Stent Placement and Removal Procedures
Description: Length of stent placement procedures and stent removal procedures.
Time Frame: Initial stent placement procedure to 24 month follow-up
Measure: Median (Full Range); unit: minutes
Units Other Than Participants: Procedures
Arm/Group | Metal Stents | Plastic Stents
Number analyzed (Participants) | 80 | 84
Number analyzed (Procedures) | 192 | 302
minutes | 26 [3 to 182] | 28 [5 to 144]
Statistical Analysis 1: Comparison: Metal Stents vs Plastic Stents; Test type: Superiority; p = .519, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Stents Placed
Description: Number of stents placed throughout study to 24 month follow-up
Time Frame: Initial stent placement procedure to 24 month follow-up
Population: Of 80 participants in metal stent arm, 1 participant never had a stent placed. Of 84 participants in plastic stent arm, 2 participants never had a stent placed, 1 participant withdrew from the study.
Measure: Mean (Standard Deviation); unit: number of stents
Arm/Group | Metal Stents | Plastic Stents
Number analyzed (Participants) | 79 | 81
number of stents | 2.3 (3.3) | 6.7 (4.4)
Statistical Analysis 1: Comparison: Metal Stents vs Plastic Stents; Test type: Superiority; p < .001, Negative binomial

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Metal Stents | Plastic Stents
All-Cause Mortality (participants affected / at risk) | 5/80 | 3/84
Serious Adverse Events (participants affected / at risk) | 19/80 | 16/84
Other Adverse Events (participants affected / at risk) | 3/80 | 8/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Metal Stents (N=80) | Plastic Stents (N=84)
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Cholangitis/fever/jaundice (Gastrointestinal disorders) | 7 | 9
Cholecystitis (Gastrointestinal disorders) | 3/69 | 1/72 — among patients with a gallbladder
Post-ERCP pancreatitis (Gastrointestinal disorders) | 2 | 0
Acute-on-chronic pancreatitis (Gastrointestinal disorders) | 2 | 0
Perforation of duodenum (Gastrointestinal disorders) | 0 | 1
Post-sphincterotomy bleed (Gastrointestinal disorders) | 1/77 | 0/76 — among patients who had a sphincterotomy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metal Stents (N=80) | Plastic Stents (N=84)
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Oedema (Gastrointestinal disorders) | 0 | 1
Acute Pancreatitis (Gastrointestinal disorders) | 0 | 1
Upper Respiratory Tract Infection (Gastrointestinal disorders) | 0 | 1
Chronic Obstruction Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-02-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT01543256/Prot_000.pdf
  • Statistical Analysis Plan (2013-03-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT01543256/SAP_001.pdf